CLINICAL TRIAL: NCT06768827
Title: Pathogenic Mechanisms of Obesity and Its Cardiometabolic Complications
Brief Title: New Mechanisms of Obesity
Acronym: NMoO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2000038988; R01DK140672 (NIH)
Record Dates: First submitted 2025-01-06; First posted 2025-01-10 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Obesity and Overweight; Insulin Resistance; Obesity and Obesity-related Medical Conditions
Keywords: Obesity; Youth; Insulin Resistance; Intestinal Fermentation
MeSH Terms: conditions — Obesity; Overweight; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remote physical exercise (Experimental)
  Interventions: Other: Lactulose Oral Product
- Control physical exercise (Active Comparator)
  Interventions: Other: Lactulose Oral Product

INTERVENTIONS:
Other: Lactulose Oral Product — Each arm will undergo a study to induce colonic fermentation through lactulose at the beginning and at the end of the 12 weeks.

SUMMARY:
Given the pervasiveness of Pediatric Obesity, it is imperative to understand its pathophysiology and develop alternative strategies to reverse this condition. Herein, investigators propose to elucidate the interaction between colonic fermentation and insulin resistance in modulating metabolism in youth with obesity.

DETAILED DESCRIPTION:
Pediatric obesity is a major health burden affecting millions of children and adolescents as it predisposes to the development of cardio-metabolic diseases early in life, such as insulin resistance, fatty liver disease and type 2 diabetes. Investigators have recently completed a series of studies to understand the relationship between the intestinal microbial activity and human metabolism in youth. It was observed that intestinal fermentation, a process through which fermentable carbohydrates are processed by intestinal bacteria, results in a variety of biological responses aimed at protecting the human body from developing obesity and some of its metabolic complications, such as insulin resistance and ectopic fat accumulation. In particular, investigators observed that intestinal fermentation causes 1- a reduction of plasma free fatty acids (FFA), due to the inhibition of adipose tissue lipolysis (ATL); 2- a marked entero-endocrine response to reduce appetite, characterized by an increase in the production of peptide YY (PYY) and glucagon-like peptide1 (GLP-1) and a reduced production of ghrelin. In addition, investigators observed that some intestinal fermentation responses are impaired in youth with obesity and insulin resistance (OIR). In light of this evidence, the current proposal will address: 1- how adipose tissue lipolysis response to intestinal fermentation is affected by insulin resistance; 2- whether changes in ATL, observed when fermentation occurs, are also associated with a reduction of glycerol derived neo-gluconeogenesis; 3- if physical activity may restore the entero-endocrine and adipose tissue response to intestinal fermentation in youth with insulin resistance. This is the first study to test the effect of insulin resistance on the relationship between intestinal microbial metabolic activity and human metabolism (namely adipose tissue lipolysis, gluconeogenesis and entero-endocrine response). The results obtained will provide fundamental insight into how insulin resistance occurring in youth with obesity affects the metabolic response to fermentable carbohydrates. In fact, despite the large body of literature showing an association between intestinal microbial fermentation and human metabolism, how and whether insulin resistance may modulate this association remains unknown.

ELIGIBILITY:
Inclusion Criteria:

* Age 15 to 22 years
* In puberty (girls and boys: Tanner stage III-V);
* BMI >85th

Exclusion Criteria:

* Pregnancy;
* endocrinopathies (e.g., Cushing syndrome);
* substance abuse;
* medications affecting insulin resistance such as metformin, GLP-1 analogues; -
* high fibers intake (> 30g/day) as assessed by a 3-day food record.

Ages: 15 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 55 (Estimated)
Dates: Start 2025-11-13 (Actual); Primary Completion 2030-03-31 (Estimated); Study Completion 2030-03-31 (Estimated)

PRIMARY OUTCOMES:
CHANGES IN ADIPOSE TISSUE LIPOLYSIS (ATL) | 6 hours
  Changes in adipose tissue lipolysis occurring after colonic fermentation (stimulated by lactulose) will be compared between youth with obesity and insulin resistance (OIR) and with obesity and without insulin resistance (OIS). Lipolysis will be measured by using change in D5-glycerol concentration.
CHANGES IN GLUCONEOGENESIS | 6 hours
  Gluconeogenesis (GLC) will be measured using change in deuterium oxide concentration after colonic fermentation due to lactulose ingestion and compared between OIS and OIR.
CHANGES IN ADIPOSE TISSUE LIPOLYSIS (ATL) | Baseline and 12 weeks
  Changes in ATL due to colonic fermentation will be measured in two groups of OIR youth. One group will undergo physical activity for 12 weeks and another group will undergo a control intervention. Lipolysis will be measured by using change in D5-glycerol concentration.

SECONDARY OUTCOMES:
CHANGES IN PEPTIDE YY (PYY) concentration | Baseline and 12 weeks
  Changes in PYY concentration after lactulose intervention will be compared between OIS and OIR.
CHANGES IN GHRELIN concentration | Baseline and 12 weeks
  Changes in GHRELIN concentration after lactulose intervention will be compared between OIS and OIR.

CONTACTS AND LOCATIONS:
Overall Officials: NICOLA SANTORO, MD, PhD, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
Published IPD will be shared at the end of the study
Supporting Information: Analytic Code
Time Frame: a year after the completion of the study
Access Criteria: Published IPD will be made available as an appendix to the paper published using the data generated through FigShare or other websites.